CLINICAL TRIAL: NCT05644782
Title: The Role of Gut-skin Axis in Psoriasis: a Randomized Placebo-controlled Dietary Approach to Assess Clinical Efficacy in Mild-to-moderate Psoriasis
Brief Title: Dietary Approach to Mild-to-moderate Psoriasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Collaborators: Aurelio Seidita (Unknown)
Responsible Party: Principal Investigator, Pasquale Mansueto, Principal Investigator, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACPM30
Record Dates: First submitted 2022-10-27; First posted 2022-12-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis; Gluten Sensitivity
Keywords: psoriasis; gluten sensitivity; gluten-free diet
MeSH Terms: conditions — Psoriasis; Celiac Disease | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled, cross-over, single center clinical trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open wheat challenge group (Active Comparator): Before starting the elimination diet (time 0, T0), intervention patients will be evaluated by experienced dermatologists, as well as by physicians with expertise in the field of food intolerance about GI and extraintestinal symptoms related to foods intake. Moreover, all these subjects will be subjected to blood, urine, and stools collections, and to a dietary consult, and a food and symptom's diary will be provided to all patients, which must be filled-in daily. After 2 months of elimination diet (time 1, T1), intervention patients will be evaluated again both clinically and by laboratory techniques, identically to T0. At this time-point, intervention patients will go to an open challenge, with reintroduction of wheat. After 2 weeks of open diet or whenever dermatologic, intestinal and/or extraintestinal symptoms should return or intensify (T2int), patients will be valued again both clinically and by laboratory techniques, identically to T0 and T1, and then will end the study.
  Interventions: Other: Open wheat challenge
- Placebo group (Placebo Comparator): Before starting the elimination diet (time 0, T0), control patients will be evaluated by experienced dermatologists, as well as by physicians with expertise in food intolerance. Moreover, patients will be subjected to blood, urine, and stools collections, and to a dietary consult, and a food and symptom's diary will be provided. After 2 months of elimination diet (time 1, T1), patients will be evaluated, identically to T0. Then, control patients will be asked to repeat the elimination diet, this time removing wheat and all cow's milk products for further 2 months (T2con). Then, patients will be valued again both clinically and by laboratory techniques, identically to T0 and T1. Then, patients will go to an open challenge, with reintroduction of wheat. After 2 weeks of open diet or whenever dermatologic, intestinal and/or extraintestinal symptoms should return or intensify (T3con), patients will be valued again, identically to T0, T1 and T2con, and then will end the study.
  Interventions: Other: Placebo challenge

INTERVENTIONS:
Other: Open wheat challenge — Patients randomized to intervention diet group will have to follow a diet with elimination of wheat and cow's milk products for 2 months; after that they will be exposed to an open wheat challenge, with reintroduction of wheat. After 2 weeks of open diet, or whenever dermatologic, intestinal and/or extraintestinal symptoms should return or intensify, all patients will be revaluated and will end the study.
  Other Names: Wheat
  Arms: Open wheat challenge group
Other: Placebo challenge — Patients randomized to control diet group will have to follow a diet with elimination of rice and turkey's meat products for 2 months; after that they will crossover to a wheat and cow's milk products free diet and, finally, after 2 months, they will be exposed to an open wheat challenge, with reintroduction of wheat. After 2 weeks of open diet, or whenever dermatologic, intestinal and/or extraintestinal symptoms should return or intensify, all patients will be revaluated and will end the study.
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
Psoriasis is a systemic chronic inflammatory immune-mediated disease whose etiopathogenetic mechanisms involve genetic predisposition, and immunological and environmental factors. Its prevalence is about 3% in adults, and it is characterized by well-demarcated, erythematous plaques, covered by silvery-white scales, in elbows, knees, trunk, and scalp. However, psoriasis is far from being considered just a dermatologic condition because the cytokine's cascade, which lays behind its inflammatory and immune-mediated pathogenesis, can determine multiple systemic manifestations. In addition, several patients with psoriasis often complains of gastrointestinal (GI) symptoms. Therefore, authors focused their attention over the gut-skin axis and its possible pathogenetic and immunoregulatory role in psoriasis (i.e., altered gut barrier, increased blood concentration of gut microbiota-derived metabolites, systemic inflammation). In this context, several dietetic approaches (e.g., Mediterranean, low calories, protein-restricted, vegetarian diets, and gluten-free diet, GFD) have shown a certain efficacy in improve psoriasis cutaneous and systemic manifestations. In recent years, the existence of a wheat-related disorder in patients who do not suffer from CD or wheat allergy (WA) has been definitively ascertained and defined as Non-Celiac Wheat Sensitivity (NCWS). Its prevalence in the general population is unknown, but self-reported NCWS is around 10%. This condition is characterized by both GI and extraintestinal symptoms, which are triggered by wheat ingestion. In these patients, wheat ingestion might lead to alteration in intestinal permeability and gut microbiota and to systemic immune activation and inflammation. Based on the evidence of gut involvement in the pathogenesis and clinical manifestation of psoriasis, as well as on the ability of gluten/wheat to increase intestinal permeability, it could be hypothesized that gluten/wheat may represents one of the pathogenetic environmental factors of psoriasis and that its intake may be able to worsen symptoms in affected patients. The investigators hypothesize that a wheat-free diet (WFD) can reduce the inflammatory state and ameliorate the clinical symptoms in psoriasis patients. The successive clinical and immunologic reaction to the re-exposure to wheat ingestion, performed by an open challenge, will be also evaluated to confirm a wheat-dependent mechanism and to understand the underlining physiopathology.

DETAILED DESCRIPTION:
Psoriasis is a systemic chronic inflammatory immune-mediated disease whose etiopathogenetic mechanisms involve genetic predisposition, as well as immunological and environmental factors. Its prevalence is about 3% in adults, and it is characterized by well-demarcated, erythematous plaques, covered by silvery-white scales, in elbows, knees, trunk, and scalp, with a typical pair distribution. However, psoriasis is far from being considered just a dermatologic condition because the cytokine's cascade [including interleukin (IL)-1β, IL-17, IL-22, IL-23, Interferon (IFN)-γ, and Tumor Necrosis Factor (TNF)-α], which lays behind its inflammatory and immune-mediated pathogenesis, can determine multiple systemic manifestations. Several reports assess that, especially in moderate-to-severe psoriasis, the same inflammatory cytokines, found in cutaneous plaques, can be found in blood, and should be considered the enhancers of a chronic inflammatory condition, which, in long-term, will flow in systemic comorbidities, such as psoriatic arthritis, cardiovascular diseases, diabetes mellitus, obesity, nonalcoholic fatty liver disease, and inflammatory bowel disease.

In addition, a variable percentage of psoriatic patients (0.2-4.3%) may present with concomitant celiac disease (CD), a well-known immune-mediated bowel disease, as well as patients suffering from CD have an increased risk of psoriasis development, and, finally, several patients with psoriasis often complains of gastrointestinal (GI) symptoms.

These evidences have recently induced authors to focus their attention over the gut-skin axis and its possible pathogenetic and immunoregulatory role in psoriasis. In this context, some studies analyzed the role of intestinal permeability and, more specifically, of the gut barrier integrity, proving that an altered gut barrier is associated with GI symptoms, systemic inflammation, and increased blood concentration of gut microbiota-derived metabolites (e.g., trimethylamine N-oxide). Confirming a strict relationship between psoriasis and gut, from a clinical point of view, several dietetic approaches (e.g., Mediterranean, low calories, protein-restricted, and vegetarian diets) have shown a certain efficacy in improve psoriasis cutaneous and systemic manifestations. Moreover, some authors showed a positive effect of a gluten-free diet (GFD) over Psoriasis Area and Severity Index (PASI) score, even if contrasting data are reported, and, to date, no large randomized controlled trials have been performed.

In recent years, the existence of a wheat-related disorder in patients who do not suffer from CD or wheat allergy (WA) has been definitively ascertained and defined as Non-Celiac Wheat Sensitivity (NCWS). Its prevalence in the general population is unknown, but self-reported NCWS is around 10%. This condition, initially named as Non-Celiac Gluten Sensitivity, assuming that, as in CD, gluten was the main culprit, is characterized by both GI [irritable bowel syndrome (IBS)-like and functional dyspepsia-like] and extraintestinal (e.g., fatigue, neuropsychiatric disorders, dermatitis, gynecological alterations, etc.) symptoms, which are triggered by wheat ingestion. Moreover, an increasing number of data have shown that patients with NCWS could have an association with autoimmune diseases, including thyroiditis, Sjogren's syndrome, undifferentiated connective tissue disease, and psoriatic arthritis. Conflicting data have been reported about the underlying physiopathology and possible symptom's triggers. Some authors identified a prevalent role for fermentable oligosaccharides-disaccharides-monosaccharides and polyols (FODMAPs), other the activation of both innate and acquired immunity. More recently, it has been shown that wheat has high concentrations of wheat amylase-trypsin inhibitors (ATIs), proteins able to activate innate immunity via toll-like receptor-4 (TLR-4) on myeloid cells. Orally ingested ATIs increase intestinal inflammation by activating gut and mesenteric lymphnode myeloid cells. A possible role in this fragmented and articulated context has been attributed to alteration of intestinal permeability. It has been known for years how exposure to gliadin, both in CD and in healthy patients (albeit with reduced levels in the latter), is able to alter intestinal permeability acting on zonulin release and signaling mechanisms. When the integrity of the intestinal barrier is compromised, penetration of toxic wheat peptides into the intestinal lamina propria could be favored, determining the onset of an inflammatory response activated by local immune system through the intervention of antigen presenting cells (APC), particularly dendritic ones. Finally, both psoriatic and NCWS patients seems to have quantitative and qualitative disbalances of gut microbiota, which could influence severity and course of these diseases. However, data on this point are conflicting and this correlation is far from being unanimously accepted.

Based on the evidence of gut involvement (i.e., influence of GFD on symptoms, increased intestinal permeability, altered microbiota) in pathogenesis and clinical manifestation of psoriasis, as well as on the ability of gluten/wheat to increase intestinal permeability, altering zonulin mechanisms of regulation and signaling, and the ability of some of its components (ATIs, but not only) to activate a local inflammatory response, it could be hypothesized that gluten/wheat may represents one of the pathogenetic environmental factors of psoriasis and that its intake may be able to worsen symptoms in affected patients.

In the investigators' hypothesis, exposure to gluten/wheat would cause a release of zonulin, which, binding to the surface of the intestinal epithelial cells, is able to modify cell cytoskeleton and cause the loss of normal occludins function, ultimately leading to an increased intestinal monolayer permeability. This increase in permeability would result in greater exposure of the immune system cells to gluten/wheat molecules via activation of TLR-4, with an increase in the infiltration and activation of myeloid cells in the intestinal mucosa and an augmented activity of lymphnode dendritic and myeloid cells. Such local inflammatory response, associated with an increase of circulating antigens coming from the gut's modified permeability, would have systemic repercussions, with alteration of normal cytokine pattern (e.g., increase of IL-1β, IL-22, IL-23, and TNF-α) and activation of plasmacytoid dendritic cells, as well as of other innate immune cells, in the skin. This background, in predisposed patients, represents the trigger for activation of myeloid dendritic cells and macrophages, IL-12, IL-23, and TNF-α-mediated recruitment of T helper type 17 (Th17) and T cytotoxic type 17 (Tc17) lymphocytes, and production of a new cytokines pattern (mainly IL-17A, and IFN-γ), which can stimulate keratinocytes to proliferate and produce antimicrobial peptides and other proinflammatory cytokines. Such complex cytokine's pattern produced by immune cells and keratinocytes, creates a positive feedback loop, perpetuating the inflammatory response which leads to clinical manifestation of psoriasis.

Therefore, the investigators hypothesize that a wheat-free diet (WFD) can reduce the inflammatory state and ameliorate the clinical symptoms in psoriatic patients. The successive clinical and immunologic reaction to the re-exposure to wheat ingestion, performed by an open challenge, will be also evaluated to confirm a wheat-dependent mechanism and to understand the underlining physiopathology.

Overall, the project results might provide data about a possible therapeutic role of a WFD in psoriasis, improve the knowledges about the relationship between intestinal permeability and systemic inflammation in psoriasis, and reveal, at least in part, the pathogenic mechanisms underlying NCWS.

Starting from the hypothesis of an altered gut-skin axis, based on altered intestinal permeability and systemic response, the investigators aim to:

1. identify the prevalence of self-reported NCWS in psoriatic patients;
2. assess the overall effect that a WFD plus cow's milk products free diet (CMPFD) determines in symptoms control and quality of life (QoL) of the patients affected with psoriasis; the investigators decided to include a CMPFD in association with a WFD because, according to several authors, including our previous studies, NCWS, and more generally gluten-related disorders, are often associated with multiple foods intolerance, first of all cow's milk products intolerance;
3. evaluate, by an open wheat challenge, the real frequency of a coexistent NCWS condition;
4. assess the possible role played by wheat ingestion in the pathogenesis and molecular mechanisms of psoriasis and NCWS by analyzing the variation of intestinal permeability and gut microbiota, in association with cytokine pattern typical of psoriasis.

ELIGIBILITY:
Inclusion criteria of psoriasis patients

* age >18 and <65 years;
* no systemic therapy for psoriasis for at least 3 months before inclusion in the study;
* negativity of anti-deamidated gliadin protein (anti-DGP) immunoglobulins (Ig) class A (IgA) and immunoglobulins (Ig)G, anti-tissue transglutaminase (anti-tTG) class IgA and IgG, and Endomysium antibodies (EmA);
* absence of WA (negative prick-test and/or specific serum immunoglobulins (Ig)E assay for wheat, gluten, and gliadin).

Exclusion criteria of psoriasis patients age <18 and >65 years;

* severe chronic plaque-type psoriasis (based on BSA);
* self-exclusion of gluten/wheat from the diet and refusal to reintroduce it, for diagnostic purposes, before entering the study;
* pregnancy;
* alcohol and/or drug abuse;
* Helicobacter pylori and other bacterial and/or parasitic infections;
* diagnosis of chronic inflammatory bowel disease and other organic pathology affecting the digestive system (e.g., severe liver disease), nervous system diseases, major psychiatric disorders, immunological deficits, and impairments that limit physical activity;
* diagnosis of cancer
* treatment with steroids and/or immunological therapies;
* patients undergoing chemotherapy and/or radiotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Self-perceived non-celiac wheat sensitivity (NCWS) questionnaire in psoriasis patients | Before enter the study.
  To identify psoriasis patients reporting a self-perceived NCWS; all patients will be asked to answer, consecutively, to a validated questionnaire for the self-assessment of wheat and other foods' intolerance. This is a questionnaire self-compiled by patients consisting of three sections: 1) general information (eg. age, sex, highest completed education level, etc.) 2) wheat-related symptoms (sore 0 = no symptoms, score = 1, symptoms after wheat intake; if score = 1 other question qualitatively inquire the symptoms evoked by wheat intake, eg. what kind of symptoms, how long patient perceive this problem, etc.); 3) other foods-related symptoms (score 0 = no symptoms, score 1 = symptoms after intake of other foods; if score = 1 other question qualitatively inquire the symptoms evoked by the intake of the specific food reported by the patients, eg. what kind of symptoms, how long patient perceive this problem, etc.)
Effect of WFD plus CMPFD in changing symptoms of psoriasis patients as assessed by BSA | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60).
  To assess the effect that a WFD plus CMPFD determines in symptoms of patients affected with psoriasis the following score will be used: Body Surface Area (BSA), representing the percentage of cutaneous area affected by psoriasis.
Effect of WFD plus CMPFD in changing symptoms of psoriasis patients as assessed by Psoriasis Area Severity Index | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60).
  To assess the effect that a WFD plus CMPFD determines in symptoms of patients affected with psoriasis the following score will be used: Psoriasis Area Severity Index (PASI), a composite evaluation for psoriasis severity, subscoring for erythema, induration, scaling, and percentage of body-surface area affected. The rating scale includes 4 levels: No Psoriasis, Mild Psoriasis, Moderate Psoriasis, and Severe Psoriasis.
Effect of WFD plus CMPFD in changing symptoms of psoriasis patients as assessed by IGA | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60).
  To assess the effect that a WFD plus CMPFD determines in symptoms of patients affected with psoriasis the following score will be used: Investigator's Global Assessment (IGA), a 5-point instrument for rating the clinician's impression of the overall severity of the psoriasis, from 0, clear skin, to 4, severe disease.
Effect of WFD plus CMPFD in changing symptoms of psoriasis patients as assessed by GSRS | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60).
  To assess the effect that a WFD plus CMPFD determines in symptoms of patients affected with psoriasis the following score will be used: Gastrointestinal Symptom Rating Scale (GSRS), assessment scale for irritable bowel syndrome-like and functional dyspepsia-like symptoms, providing for a score ranging from 15 to 60).
Effect of WFD plus CMPFD in changing symptoms of psoriasis patients as assessed by Extraintestinal symptoms rating scale. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60).
  To assess the effect that a WFD plus CMPFD determines in symptoms of patients affected with psoriasis the following score will be used: Extraintestinal symptoms rating scale, a scoring system based on the symptoms most frequently observed in NCWS patients, providing for a score ranging from 9 to 34.
Effect of WFD plus CMPFD in changing Quality of Life (QoL) of psoriasis patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60).
  To assess the effect that a WFD plus CMPFD determines in QoL of patients affected with psoriasis, both of the intervention and the control group. The following score will be used: Dermatology Life Quality Index (DLQI, a validated instrument to evaluate quality of life for skin disease, providing for a score ranging from 0 to 30 points, with higher scores indicating a greater effect on quality of life).

SECONDARY OUTCOMES:
Effect of open wheat challenge in symptoms changing of psoriasis patients as assessed by BSA | Day 60; 2 weeks of open wheat challenge (Day 75).
  To evaluate, by an open wheat challenge, the frequency of a coexistent NCWS condition in psoriasis patients, both of the intervention group (T2int) and the control group (T3con). The following score will be used: Body Surface Area (BSA), representing the percentage of cutaneous area affected by psoriasis.
Effect of open wheat challenge in symptoms changing of psoriasis patients as assessed by Psoriasis Area Severity Index | Day 60; 2 weeks of open wheat challenge (Day 75).
  To evaluate, by an open wheat challenge, the frequency of a coexistent NCWS condition in psoriasis patients, both of the intervention group (T2int) and the control group (T3con). the following score will be used: Psoriasis Area Severity Index (PASI), a composite evaluation for psoriasis severity, subscoring for erythema, induration, scaling, and percentage of body-surface area affected. The rating scale includes 4 levels: No Psoriasis, Mild Psoriasis, Moderate Psoriasis, and Severe Psoriasis.
Effect of open wheat challenge in symptoms changing of psoriasis patients as assessed by IGA. | Day 60; 2 weeks of open wheat challenge (Day 75).
  To evaluate, by an open wheat challenge, the frequency of a coexistent NCWS condition in psoriasis patients, both of the intervention group (T2int) and the control group (T3con). The following score will be used: Investigator's Global Assessment (IGA), a 5-point instrument for rating the clinician's impression of the overall severity of the psoriasis, from 0, clear skin, to 4, severe disease.
Effect of open wheat challenge in symptoms changing of psoriasis patients as assessed by GSRS. | Day 60; 2 weeks of open wheat challenge (Day 75).
  To evaluate, by an open wheat challenge, the frequency of a coexistent NCWS condition in psoriasis patients, both of the intervention group (T2int) and the control group (T3con).The following score will be used: Gastrointestinal Symptom Rating Scale (GSRS), assessment scale for irritable bowel syndrome-like and functional dyspepsia-like symptoms, providing for a score ranging from 15 to 60).
Effect of open wheat challenge in symptoms changing of psoriasis patients as assessed by Extraintestinal symptoms rating scale. | Day 60; 2 weeks of open wheat challenge (Day 75).
  To evaluate, by an open wheat challenge, the frequency of a coexistent NCWS condition in psoriasis patients, both of the intervention group (T2int) and the control group (T3con). The following score will be used: Extraintestinal symptoms rating scale, a scoring system based on the symptoms most frequently observed in NCWS patients, providing for a score ranging from 9 to 34.
Effect of open wheat challenge in Quality of Life (QoL) changing of psoriasis patients. | Day 60; 2 weeks of open wheat challenge (Day 75).
  To assess the effect that an open wheat challenge determines in QoL of patients affected with psoriasis, both of the intervention (T2int) and the control group (T3con). The following score will be used: DLQI (a validated instrument to evaluate quality of life for skin disease, providing for a score ranging from 0 to 30 points, with higher scores indicating a greater effect on quality of life).
Erythrocyte sedimentation rate (ESR) changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Laboratory blood analysis will be performed to assess erythrocyte sedimentation rate (ESR)
C-reactive protein (CRP) changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Laboratory blood analysis will be performed to assess C-reactive protein (CRP)
Complete blood count changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Laboratory blood analysis will be performed to assess complete blood count
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interleukin (IL)-1β
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interleukin (IL)-2
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interleukin (IL)-4
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interleukin (IL)-5
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interleukin (IL)-6
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interleukin (IL)-8
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interleukin (IL)-10
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interleukin (IL)-17A
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interleukin (IL)-22
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interleukin (IL)-23,
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: Tumor Necrosis Factor (TNF)-α
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: interferon (IFN)-γ
Peripheral blood ELISA analysis of inflammatory cytokines changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of inflammatory cytokines pattern will be performed to assess: Toll-Like Receptor (TLR)-4.
Peripheral blood cytofluorimetric analysis to evaluate expression of lymphocytes typical of psoriasis | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood cytofluorimetric analysis will be performed to assess expression of lymphocytes typical of psoriasis pathogenetic pattern [i.e., T helper (Th)17, and T cytotoxic (Tc)17].
Peripheral blood ELISA analysis of intestinal permeability markers changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of intestinal permeability markers will be performed to assess: zonulin
Peripheral blood ELISA analysis of intestinal permeability markers changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of intestinal permeability markers will be performed to assess: F-Actin
Peripheral blood ELISA analysis of intestinal permeability markers changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of intestinal permeability markers will be performed to assess: intestinal fatty acid-binding protein (i-FABP)
Peripheral blood ELISA analysis of intestinal permeability markers changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of intestinal permeability markers will be performed to assess: lipopolysaccharide (LPS)
Peripheral blood ELISA analysis of intestinal permeability markers changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Peripheral blood ELISA analysis of intestinal permeability markers will be performed to assess: LPS-binding protein (LBP)
Lactulose(LA)/Mannitol(MA) test changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  LA/MA test will be performed to assess in vivo intestinal permeability.
Fecal ELISA analysis of inflammatory gut marker changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Fecal ELISA analysis of inflammatory gut marker will be performed to assess fecal calprotectin.
Gut microbiota changing in psoriasis and NCWS patients. | Start of the study (Day 0); 2 months of wheat elimination diet (Day 60); 2 weeks of open wheat challenge (Day 75)
  Gut microbiota assessment will be performed by analysis and quantification of gut microbioma on stools samples. After fecal collection, bacterial DNA will be extracted by cetyltrimethyl ammonium bromide. A simple and inexpensive physical lysis method for DNA and RNA extraction from freshwater microalgae and 16S ribosomal ribonucleic acid (rRNA) sequencing will be performed by polymerase chain reaction (PCR) methods, using universal primers. The resulting fragments will be then sequenced by pyrosequencing. Each reading will be compared with a database of known 16S rRNA sequences, using the BLAT program by phylogenetically assigning the most specific and reliable nodes. This method of assigning the obtained data leads to a "weighted" phylogenetic tree that characterizes well the bacterial content of the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, Study Director — University of Palermo; Maria R. Bongiorno, MD, Study Chair — University of Palermo
Locations (3):
- Italy (3):
  - Dermatology Department of the University Hospital 'P. Giaccone' of Palermo, Italy,, Palermo, Palermo
  - Internal Medicine Department of the University Hospital of Palermo, Palermo, Palermo
  - Internal Medicine Division of the "Cervello-Villa Sofia" Hospital, Palermo, PA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marsili F, Travaglini M, Stinco G, Manzoni R, Tiberio R, Prignano F, Mazzotta A, Cannavo SP, Cuccia A, Germino M, Bongiorno MR, Persechino S, Florio T, Pettinato M, Tabanelli M, Sarkar R, Aloisi E, Bartezaghi M, Orsenigo R. Effectiveness of cyclosporine A in patients with moderate to severe plaque psoriasis in a real-life clinical setting in Italy: the TRANSITION study. J Dermatolog Treat. 2022 Feb;33(1):401-407. doi: 10.1080/09546634.2020.1757017. Epub 2020 Apr 30. PMID 32349568
- [Result] Pistone G, Gurreri R, Tilotta G, Caruso P, Curiale S, Bongiorno MR. Timing of quality of life improvements in psoriatic patients treated with different systemic therapies. Dermatol Ther. 2019 Sep;32(5):e13021. doi: 10.1111/dth.13021. Epub 2019 Jul 31. PMID 31306540
- [Result] Carroccio A, Giambalvo O, Blasca F, Iacobucci R, D'Alcamo A, Mansueto P. Self-Reported Non-Celiac Wheat Sensitivity in High School Students: Demographic and Clinical Characteristics. Nutrients. 2017 Jul 19;9(7):771. doi: 10.3390/nu9070771. PMID 28753927
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366